CLINICAL TRIAL: NCT06231602
Title: The Relationship Between Maternal Perinatal Depression and Feeding Behavior Among Primiparas
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202310157RINC
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Perinatal Depression; Breastfeeding; Complementary Feeding
Keywords: prenatal depression; postpartum depression; breastfeeding; complementary feeding
MeSH Terms: conditions — Breast Feeding; Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to explore the impact of pregnancy depression on infant feeding, and to explore the two-way relationship between postpartum depression and infant feeding. Participants will be asked to finish questionnaires four times (24 weeks of pregnancy to before delivery, 2 month postpartum, 4 month postpartum, 6 month postpartum).

DETAILED DESCRIPTION:
Background: Perinatal depression and infant feeding (breastfeeding and complementary feeding) are important global health issues. The prevalence of perinatal depression is high around the world, and breastfeeding rates in middle- and high-income countries are on a downward trend. Past research has pointed out that perinatal depression is related to infant feeding. However, there is a lack of research on the impact of maternal depression on infant feeding in Asian Chinese pregnant women, and "whether there is a bidirectional causal relationship between postpartum depression and infant feeding" remains unclear.

Purpose: To explore the impact of pregnancy depression on infant feeding, and to explore the two-way relationship between postpartum depression and infant feeding.

Method: This is a longitudinal cohort study. It's estimated to recruit 500 pregnant women. It is planned to recruit participants at the Obstetrics and Gynecology Clinic of National Taiwan University Hospital. At the same time, research recruitment advertisements will also be posted online. This study will collect data by questionnaires distributed a total four times (24 weeks of pregnancy to before delivery, 2 month postpartum, 4 month postpartum, 6 month postpartum). Variables include: sociodemographics, maternal variables (parity, number of births, planned pregnancy, maternal complications, mode of delivery, height and weight during pregnancy and postpartum, blood pressure), infant variables (gender, health status , height, weight), anticipatory feeding schedule, health-risk behaviors (smoking and alcohol use), social support, situation of breastfeeding and complementary feeding, reactive feeding, sleep, fatigue, exercise habits, and tendency to depression.

ELIGIBILITY:
Inclusion Criteria:

* Primipara
* Adult women over 18 years old
* Those with no recurrent pregnancy loss and stable signs of pregnancy
* Those who agree to participate in this study

Exclusion Criteria:

* No exclusion conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The participants of this study are pregnant women because this study aims to explore the impact of pregnancy depression on infant feeding, and to explore the two-way relationship between postpartum depression and infant feeding.
Study Population: It is planned to recruit participants at the Obstetrics and Gynecology Clinic of National Taiwan University Hospital. At the same time, research recruitment advertisements will also be posted online.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
maternal variables | 24 weeks of pregnancy to before delivery, 2 month postpartum, 4 month postpartum, 6 month postpartum
  Questions contain parity, number of births, planned pregnancy, maternal complications, mode of delivery, height in centimeters, weight in kilograms, blood pressure, etc. Height and weight will be measured during pregnancy and postpartum(Height and weight will be combined to report BMI in kg/m^2).
infant variables | 2 month postpartum, 4 month postpartum, 6 month postpartum
  Questions contain gender, health status , height in centimeters, weight in grams.
perinatal depression | 24 weeks of pregnancy to before delivery, 2 month postpartum, 4 month postpartum, 6 month postpartum
  Depression was measured using the Edinburgh Postnatal Depression Scale.
breastfeeding situation | 2 month postpartum, 4 month postpartum, 6 month postpartum
  Questions contain whether breastfeeding is continued, the type of feeding (breastfeeding or formula feeding), whether additional liquids are fed and the amount of feeding, etc.
complementary feeding situation | 4 month postpartum, 6 month postpartum
  Questions contain types of food, starting age of introduction, daily feeding amount and daily feeding times, etc.

CONTACTS AND LOCATIONS:
Overall Officials: HUNG-HUI CHEN, Principal Investigator — National Taiwan University Hostiptal
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No